CLINICAL TRIAL: NCT04648280
Title: A Multicenter, Open-label, Single-arm Trial to Evaluate the Safety, Pharmacokinetics and Antiviral Activity of Fostemsavir in Combination With Optimized Background Therapy (OBT) in HIV-1 Infected Children and Adolescents Who Are Failing Their Current Combination Antiretroviral Therapy (cART) and Have Dual- or Triple-class Antiretroviral (ARV) Resistance
Brief Title: Safety and Pharmacokinetics Evaluation of Fostemsavir + (OBT) in HIV-1 Infected Children and Adolescents Who Are Failing Their cART and Have Dual- or Triple-class Antiretroviral Resistance
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: PENTA Foundation (Network)
Collaborators: ViiV Healthcare (Industry); PHPT Foundation (Unknown); Hospital Universitario 12 de Octubre (Other); Cromsource (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHIELD (Penta22)
Record Dates: First submitted 2020-11-10; First posted 2020-12-01 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: HIV Infections With Multi Drug Resistant Virus
MeSH Terms: interventions — fostemsavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Fostemsavir (Experimental): Fostemsavir in combination with optimized background therapy (OBT) in HIV-1 infected children and adolescents who are failing their current combination antiretroviral therapy (cART) and have dual- or triple-class ARV resistance
  Interventions: Drug: Fostemsavir

INTERVENTIONS:
Drug: Fostemsavir — fostemsavir in combination with optimized background therapy (OBT) in HIV-1 infected children and adolescents who are failing their current combination antiretroviral therapy (cART) and have dual- or triple-class ARV resistance

SUMMARY:
In the SHIELD study, the study sponsor seeks to assess safety, PK and antiviral activity for children and adolescents with dual or triple class resistance. It will also assess the acceptability and swallowability of formulation among the pediatric population. The dose selection of FTR for children and adolescents ≥20kg utilized a population pharmacokinetic (POP PK) model-based approach to achieve similar adult TMR exposures following FTR 600mg BID administration with combination therapy that was demonstrated to be safe and effective in the FTR Phase 3 BRIGHTE study in HTE patients.

ELIGIBILITY:
Inclusion Criteria:

* Male and female HIV-1 infected paediatric participants from 6 years old and weighing at least 20 kg to less than 18 years of age.
* Antiretroviral-experienced with documented historical or baseline resistance to one or more agents in at least two classes. All resistance has to be properly documented.
* Failing current antiretroviral regimen with a confirmed plasma HIV-1 RNA ≥ 1000 c/mL (first value from Investigator within 6 months of screening visit, with the second value obtained from Screening labs, without a decline greater than 1 log10, and no value <1000 in between).
* Documented resistance to at least one component of the current failing regimen per screening resistance testing.
* Must have at least 1 fully active and available agent in 2 or more ARV classes, based on current and/or documented historical resistance testing, taking into account tolerability, and other safety concerns. At least two fully active agents must be a part of the initial OBT to be paired with FTR.
* Girls who have reached menarche must have a negative pregnancy test at screening, not be breastfeeding, and be willing to adhere to effective methods of contraception if sexually active. All participants (male or female) have to agree with recommendations for effective contraception.

Exclusion Criteria:

Medical History and Concurrent Diseases:

* Unable to comply with dosing requirements (to swallow solid pharmaceutical form of the investigational medicinal product)
* Unable to comply with study visits
* Presence of a malabsorption syndrome or other gastrointestinal dysfunction which might interfere with drug absorption or render the participant unable to take oral medication.
* Any clinical condition (including but not limited to recreational drug use) or prior therapy that, in the opinion of the Investigator, would make the participant unsuitable for the study
* Pregnancy and breastfeeding

Physical and Laboratory Test Findings:

* Chronic untreated Hepatitis B virus (HBV) (however, participants with chronic treated HBV or spontaneously remitted HBV are eligible)
* HIV-2 infection
* Alanine aminotransferase (ALT) ≥5 times the upper limit of normal (ULN), OR ALT ≥3xULN and bilirubin ≥1.5xULN (with>35% direct bilirubin)
* History of unstable liver disease, decompensated cirrhosis, or known biliary disorder
* History of congestive heart failure, or congenital/acquired prolonged QT syndrome/other cardiac diseases predisposing to prolonged QTc
* Hemoglobin < 8.0 g/dL
* Platelets < 50,000 cells/mm3
* Confirmed QTcF value > 450 msec, regardless of sex, at Screening or Day 1
* Current (defined as taking the medication within 14 days of Day 1) or anticipated treatment with medication considered prohibited or restricted as per Appendix II. Certain medication will be carefully evaluated as acceptable, see Appendix II.
* Participation in an experimental drug and/or HIV-1 vaccine trial(s) within the previous 30 days
* Child in governmental care, e.g. child is a ward of the state. Note: This criterion does not apply if the child is officially adopted by a family/guardian.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2022-06-30 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Occurrence of the following events through Week 24 | 24 weeks
AUC(0-tau) | at week 1, 4, 12, 24, 48
Cmax | at week 1, 4, 12, 24, 48
Ctau of temsavir across weight bands | at week 1, 4, 12, 24, 48

SECONDARY OUTCOMES:
Proportion of patients with HIV-1 RNA <50 copies/mL | at 24 weeks and 48 weeks
  To evaluate the antiviral activity of fostemsavir + OBT
Change in log10 HIV-1 RNA from baseline | at 24 weeks and 48 weeks
Occurrence of: AEs, treatment-related AEs, AEs of Grade 3 or higher, serious AEs, and AEs leading to premature study treatment discontinuation. | at Week 48 and at the end of Study
Occurrence of WHO 3 or 4 defining events, or death | up to 156 weeks
efficacy of fostemsavir plus OBT | up to 156 weeks
  changes from baseline in CD4+ T cell counts and the percentage of CD4 + T-cells
Emergence of genotypic or phenotypic resistance to Temsavir and components of OBT | up to 156 weeks

CONTACTS AND LOCATIONS:
Locations (10):
- United States (2):
  - The George Washington University, Children's National Health System, Washington D.C., District of Columbia
  - Children's Healthcare of Atlanta, Atlanta, Georgia
- Brazil (2):
  - Hospital Geral de Nova Iguaçu, Nova Iguaçu
  - Hospital Federal dos Servidores do Estado, Rio de Janeiro
- South Africa (6):
  - FAM-CRU, Cape Town
  - King Edward VIII Hospital, Durban
  - Rahima Moosa Mother and Child Hospital, Johannesburg
  - Wits Reproductive Health and HIV Institutel, Johannesburg
  - Kalafong Hospital, Pretoria
  - PHRU, Soweto

IPD SHARING:
Plan to Share IPD: No